CLINICAL TRIAL: NCT03177590
Title: Recording Facial and Vocal Emotional Productions in Children With Autism as Part of the JEMImE Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-HPNCL-02
Record Dates: First submitted 2017-02-22; First posted 2017-06-06 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Autism; Pervasive Developmental Disorder
Keywords: autism; Pervasive Developmental Disorder
MeSH Terms: conditions — Autistic Disorder; Child Development Disorders, Pervasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recordings of facial and vocal emotional (Experimental): Recordings of facial and vocal emotional productions during Children are performing three tasks
  Interventions: Other: Recordings of facial and vocal emotional productions

INTERVENTIONS:
Other: Recordings of facial and vocal emotional productions — Children are asked to perform three tasks:
  1. an emotional production on imitation (the child with autism or TED will imitate the emotion expressed by an animated avatar)
  2. an emotional production by mime of the emotion on command (oral and written) without visualizing the model of imitation
  3. Emotional production in context: the child with autism or EFD will describe images forming the story of Frog and as it is read, will produce the appropriate facial and vocal emotions in the context.

SUMMARY:
The purpose of the JEMImE project is to create a serious game to help children with Autism and Pervasive Developmental Disorder (PDD) develop facial and vocal emotions in context.

The objective of this study is to record facial and vocal emotional productions in children with autism and PDD in order to create an algorithm for the recognition of facial emotional expressions implemented in the serious game JEMImE.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism and Pervasive developmental disorder according to Diagnostic and Statistical Manual of Mental Disorders IV (DSM IV) criteria using scales (Autism Diagnostic Interview ADI and / or Autism Diagnostic Observation Schedule ADOS).
* Intelligence Quotient (IQ) = /> 70 (Wechsler Intelligence Scale for Children WISC IV)
* Subjects and holders of parental authority who have given their informed and written consent
* Subjects affiliated to social security system.

Exclusion Criteria:

* Subjects non affiliated to social security system.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2016-05-10 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Record facial and vocal emotional productions of children of an imitation situation | At baseline
  The outcome is the record with a 3D camera in test situations an imitation (facial and facial / vocal) situation of emotion expressed by an animated (on-screen) avatar with assessment of emotional production

SECONDARY OUTCOMES:
Record facial and vocal emotional productions of children in a situation of mime on written request | At baseline
  The outcome is the record with a 3D camera in a situation of mime (facial and facial / vocal) on written request (on screen) with assessment of emotional production
Record facial and vocal emotional productions of children in a situation of mime on presentation of an image | At baseline
  The outcome is the record with a 3D camera in a situation of mime of an emotion on presentation of an image with assessment of emotional production

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie SERRET, MD, Principal Investigator — Fondation Lenval Hôpitaux Pédiatriques de Nice CHU-LENVAL
Locations (2):
- France (2):
  - Fondation Lenval Hôpitaux Pédiatriques de Nice CHU-LENVAL, Nice
  - Hôpital de La Salpétrière - APHP, Paris

IPD SHARING:
Plan to Share IPD: No